CLINICAL TRIAL: NCT02535650
Title: An Open Label Phase II Study of Tipifarnib in Patients With Previously-Treated, Advanced, HRAS Mutant Urothelial Carcinoma
Brief Title: Study of Tipifarnib in Patients With Previously-Treated, Advanced, HRAS Mutant Urothelial Carcinoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Park, Se-Hoon, Clinical Professor, Samsung Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2015-05-039
Record Dates: First submitted 2015-08-25; First posted 2015-08-28 (Estimated); Last update posted 2022-03-08 (Actual); Status verified 2022-03

CONDITIONS: Urothelial Carcinoma
MeSH Terms: conditions — Carcinoma, Transitional Cell | interventions — tipifarnib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- tipifarnib (Experimental): Tipifarnib will be administered at a starting dose of 900 mg, po, bid on days 1-7 and 15-21 of 28-day treatment cycles.
  Interventions: Drug: tipifarnib

INTERVENTIONS:
Drug: tipifarnib — Tipifarnib will be administered at a starting dose of 900 mg, po, bid on days 1-7 and 15-21 of 28-day treatment cycles. In the absence of unmanageable toxicities, subjects may continue to receive tipifarnib treatment for up to 12 months as long as the Investigator considers that the treatment is providing clinical benefit.

SUMMARY:
Platinum-based chemotherapy is now regarded a standard first-line treatment for patients with advanced urothelial carcinoma (UC). However, patients who failed to response or experienced progression after platinum-based chemotherapy have a grim prognosis and a standard salvage treatment is not available.

UC is known to harbor multiple mutations. In the investigators' own high-throughput molecular profiling study, the most commonly observed mutations included TP53, FGFR3(fibroblast growth factor receptor 3 ) and HRAS. Since RAS signaling can be attenuated using selective farnesyl transferase (FTase) inhibitors, tipifarnib, a highly potent and selective inhibitor of FTase, was proposed to be an effective therapeutic approach in the treatment of UC.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is at least 20 years of age.
2. Subject has a histologically or cytologically confirmed diagnosis of urothelial carcinoma arising from urinary bladder or upper urinary tract.
3. Subject has been treated with platinum-based chemotherapy for advanced disease. They must have refractory or progressive disease for which there is no further curative therapy available.
4. Subject has been treated with platinum-based chemotherapy for advanced disease. They must have refractory or progressive disease for which there is no further curative therapy available.

   Subject has a tumor that carries a missense HRAS mutation according to a standard methodology using Illumina HiSeqTM. (missence non-synonymous HRAS mutation and/or STK11: rs2075606 (T>C))HRAS status may have been assessed either in primary tumor tissue, recurrent or metastatic disease.
5. Subject has consented to provide at least 10 unstained tumor slides for retrospective testing of HRAS gene tumor status.
6. Must have a life expectancy of 3 months or more
7. Subject has measurable disease according to RECIST(Response Evaluation Criteria in Solid Tumors ) v1.1 and has relapsed (progressive disease) or is refractory to prior therapy.
8. At least 2 weeks since the last systemic therapy regimen prior to enrolment. Subjects must have recovered to NCI CTCAE v. 4.03 < Grade 2 from all acute toxicities (excluding Grade 2 toxicities that are not considered a safety risk by the Sponsor and Investigator) or toxicity must be deemed irreversible by the Investigator.
9. At least 2 weeks since last radiotherapy if radiation was localized to the only site of measurable disease, unless there is documentation of disease progression of the irradiated site. Patients must have recovered from all acute toxicities from radiotherapy.
10. ECOG(Eastern Cooperative Oncology Group ) performance status of 0 or 1.
11. Acceptable liver function:

    1. Bilirubin ≤ 1.5 times upper limit of normal (x ULN); does not apply to subjects with Gilbert's syndrome diagnosed as per institutional guidelines.
    2. AST (SGOT,aspartate aminotransferase ) and ALT (SGPT,Alanine aminotransferase) ≤ 3 x ULN; if liver metastases are present, then ≤ 5 x ULN is allowed.
12. Acceptable renal function with serum creatinine ≤ 1.5 x ULN or a calculated creatinine clearance ≥ 60 mL/min using the Cockcroft-Gault or MDRD(Modification of Diet in Renal Disease ) formulas. Serum potassium with normal or ≤ CTCAE Grade 1 with or without supplementation.
13. Acceptable hematologic status (without growth factor support or transfusion dependency):

    1. ANC(absolute neutrophil count )>1500 cells/μL.
    2. Platelet count >100,000/μL.
    3. Hemoglobin >9.0 g/dL.
14. Female subjects must be either:

    1. Of non-child-bearing potential (surgically sterilized or at least 2 years post-menopausal); or
    2. If of child-bearing potential, subject must use an adequate method of contraception consisting of two-barrier method or one barrier method with a spermicide or intrauterine device. Both females and male subjects with female partners of child-bearing potential must agree to use an adequate method of contraception for 2 weeks prior to screening, during, and at least 4 weeks after last dose of trial medication. Female subjects must have a negative serum or urine pregnancy test within 72 hours prior to start of trial medication.
    3. Not breast feeding at any time during the study.
15. Written and voluntary informed consent understood, signed and dated.

Exclusion Criteria:

1. Ongoing treatment with an anticancer agent not contemplated in this protocol.
2. Prior treatment (at least 1 full treatment cycle) with an FTase inhibitor.
3. Any history of clinically relevant coronary artery disease or myocardial infarction within the last 3 years, New York Heart Association (NYHA) grade III or greater congestive heart failure, cerebrovascular attack within the prior year, or current serious cardiac arrhythmia requiring medication except atrial fibrillation.
4. Known uncontrolled brain, leptomeningeal or epidural metastases (unless treated and well controlled for at least 4 weeks prior to Cycle 1 Day 1). Subjects that develop brain metastasis during the study may have their treatment interrupted to receive a course of cranial radiation and restart trial medication after a recovery period of at least 1 week. High dose corticosteroids may be employed for the management of cranial radiation but must be tapered off before resuming treatment.
5. Non-tolerable > Grade 2 neuropathy or evidence of unstable neurological symptoms within 4 weeks of Cycle 1 Day 1.
6. Major surgery, other than diagnostic surgery, within 4 weeks prior to Cycle 1 Day 1, without complete recovery.
7. Double primary cancer of other site(s), except for cured ones at the discretion of investigator
8. Active, uncontrolled bacterial, viral, or fungal infections, requiring systemic therapy. Known infection with HIV, or an active infection with hepatitis B or hepatitis C.
9. Subjects who have exhibited allergic reactions to tipifarnib, structural compounds similar to tipifarnib or to its excipients.
10. Concomitant disease or condition that could interfere with the conduct of the study, or that would, in the opinion of the Investigator, pose an unacceptable risk to the subject in this study.
11. The subject has legal incapacity or limited legal capacity.
12. Dementia or significantly altered mental status that would limit the understanding or rendering of informed consent and compliance with the requirements of this protocol. Unwillingness or inability to comply with the study protocol for any reason.
13. QTcF interval ≥ 470 msecs

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2015-11-12 (Actual); Primary Completion 2022-03 (Estimated); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
6-month progression-free survival | Up to 6 months for each subject

SECONDARY OUTCOMES:
Duration of response | Up to 12 months for each subject
Overall survival | Until the date of death from any cause, whichever came first, assessed up to 1 year 6 months.
Safety and Tolerability | Up to 12 months for each subject
  Number of Participants With Treatment-Related Adverse Events as Assessed by CTCAE v4.0(Common Toxicity Criteria for Adverse Effects )

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung Medical Center, Seoul, South Korea